CLINICAL TRIAL: NCT05453058
Title: TALISMAN - Tracking Longitudinal Changes in MSA - International Natural History Study
Brief Title: Observational Study in Multiple System Atrophy
Acronym: TALISMAN
Status: Active, not recruiting | Type: Observational
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: 20058N
Record Dates: First submitted 2022-06-16; First posted 2022-07-12 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Multiple System Atrophy
MeSH Terms: conditions — Multiple System Atrophy | interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with possible or probable MSA: This protocol does not mandate the use of any treatments. No study medication will be administered as part of study participation. Any treatment that study patients receive will be prescribed according to the recommendations given in the local SmPCs.
  Interventions: Diagnostic Test: plasma NfL and brain MRI (vMRI, DTI, and ASL [if feasible]) only for the EU cohort

INTERVENTIONS:
Diagnostic Test: plasma NfL and brain MRI (vMRI, DTI, and ASL [if feasible]) only for the EU cohort — Biomarker assessments are mandated in this protocol (i.e., they are not expected to be done as part of routine clinical practice).
  These assessments will be conducted within the same time window as the observational assessments (at approx. 6-month intervals) and are mandated by protocol if not conducted as per clinical practice.

SUMMARY:
Talisman is global clinical study (20058N) in Multiple System Atrophy (MSA) patients. It will be conducted in two regions (China and the European Union [EU]). There will be common study objectives between China and EU regions (including prospective assessments for MSA disease progression during routine clinical visits for MSA), and this will allow for data (on common objectives) to be presented overall and stratified by region. There will also be study objectives specific to each region: 1) the clinical assessment for MSA (Unified MSA Rating Scale [UMSARS]) has not been validated using standardised methods in China, and so the psychometric properties of the Chinese version of the UMSARS will be examined in Chinese patients in this study; 2) there will be retrospective assessments and prospective protocol-mandated assessments (of Magnetic Resonance Imaging [MRI] and bloods biomarkers) and study visits for EU patients.

Because some study objectives are the same for China and the EU (i.e., prospective assessments during routine clinical visits for MSA), and other objectives are specific to each region, there will be one regional protocol for China and one regional protocol for the EU; each describing the study assessments relevant to each region.

DETAILED DESCRIPTION:
Multiple system atrophy (MSA) is a sporadic, rapidly progressing neurodegenerative disorder. Most MSA patients are diagnosed between 50 to 60 years of age and the mean survival time is 6 to 10 years from symptom onset, with few surviving more than 15 years from symptom onset. The rapid progression and complexity of the disease, as well as its unresponsiveness to drugs, such as Levodopa for parkinsonian symptoms, makes MSA a challenging disease to treat. Based on the predominant motor features at the time of clinical evaluation, MSA is classified as either MSA with predominant parkinsonism (MSA-P) or MSA with predominant cerebellar ataxia (MSA-C).

MSA is an orphan and rare disease. The prevalence estimate of MSA is 3 to 5 per 100,000 in the general population. The prevalence estimate ranges from 2 to 5 per 100,000 in the United States and European Union (EU) and from 7 to 20 per 100,000 in Japan. MSA-P comprises approximately 70% of cases in the US and EU, whilst MSA-C comprises approximately 70% of cases in Japan.

Blood and MRI biomarkers have been evaluated in MSA patients. NfL (Neurofilament light protein) levels are increased in the cerebrospinal fluid (CSF) and plasma of patients with MSA and correlate with MSA disease severity, as measured by the unified MSA rating scale (UMSARS). An accurate estimate of NfL levels over time could help monitor MSA prognosis and help define the timepoints that could be targeted for effective treatment.

Furthermore, MSA patients with abnormal brain MRI findings have faster clinical progression of MSA, as evaluated with the UMSARS total score and UMSARS Part II (clinical examination). A recent review on the role of MRI in MSA noted that whilst MRI is a promising tool for diagnosing and monitoring disease progression; well-designed, large, prospective studies are needed before MRI biomarkers could be incorporated into a neuroimaging-supported diagnosis of MSA. The knowledge gained from this study should help improve understanding of biomarkers and other disease progression outcomes in MSA. This could allow MSA disease progression to be monitored and therefore treated more effectively. Insights into the natural course of disease in MSA patients in the EU will be combined and compared with data on the natural course of disease in MSA patients in China, as part of a larger global cohort. Specifically, the natural course of MSA will be explored in patients in China (using [Chinese versions of] the same prospective observational assessments as the current prospective protocol in the EU). This will allow for data collected prospectively during routine visits for MSA in China to be combined and compared with data collected prospectively during routine visits for MSA in the EU.

The extension part of Talisman:

The extension of Talisman will describe early MSA disease progression and mortality assessed remotely via telephone call with either the participant or care-partner in 6-month intervals up until 60 months after enrolling in extension study. The long-term extension will generate knowledge on long-term disease progression and survival in MSA.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be aged between ≥40 and ≤75 years, at baseline.
2. The patient must be diagnosed with possible or probable MSA of the parkinsonian subtype (MSA-P) or cerebellar subtype (MSA-C), according to the Gilman criteria (version 2).
3. The patient must have an anticipated survival of at least 3 years in the opinion of the study investigator, at baseline.
4. The patient had onset of motor MSA symptoms within 5 years prior to the baseline visit in the judgement of the study investigator.
5. The patient must have an UMSARS Part I score of ≤16 (omitting question 11 on sexual function), at baseline.
6. The patient must have normal cognition (i.e., Montreal Cognitive Assessment [MoCA] score ≥22), at baseline.
7. The patient's caregiver must have approximately 3 hours per week contact with the patient and be available and able to accompany the patient to routine clinical visits throughout the study, to provide information on the patient's functional abilities.
8. The patient/patient's legally acceptable representative, and the patient's caregiver are willing to provide written voluntary informed consent.
9. The patient's treatments are prescribed according to routine clinical practice and local guidelines/regulations.

Exclusion criteria:

1. The patient has evidence (clinical or on MRI) and/or history of any serious neurological disorder, other intracranial or systemic diseases or conditions resulting in a diagnosis other than MSA.
2. The patient has two or more blood relatives with a history of MSA.
3. The patient is, in the investigator's opinion, unlikely to comply with the protocol.
4. The patient has previously been enroled in this study.
5. The patient is a member of the study personnel or of their immediate family or is a subordinate (or immediate family member of a subordinate) to any of the study personnel.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 140 patients with relatively early MSA from China and EU are expected to be enroled in this study during a 9-month enrolment.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-06-25 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2031-05-30 (Estimated)

PRIMARY OUTCOMES:
To describe early MSA disease progression changes in 6-month intervals over 12-months (i.e., baseline, 6-months, 12-months) | baseline, 6 months, 12 months
  Disease progression will be assessed using the Unified MSA Rating Scale (UMSARS) Part I and II (scores ranging from 0-104); higher scores indicate greater impairment
Changes from baseline to approx. 6-months after baseline and approx.12- months after baseline in plasma NfL concentrations. | baseline, 6 months, 12 months
Percentage change in brain volume in brain regions-of-interest (ROIs), as measured by volumetric MRI (vMRI). | baseline, 6 months, 12 months
Percentage change in tissue integrity in ROIs, as measured by diffusion-tensor imaging (DTI) MRI. | baseline, 6 months, 12 months

SECONDARY OUTCOMES:
To evaluate changes from baseline on the impact of disease progression on the quality of life (QoL) of the patient at 6 and 12 months | baseline, 6 months, 12 months
  Patient QoL will be measured by the European Quality of Life Five Dimensions questionnaire 5 level version (EQ-5D-5L)
To evaluate changes from baseline on the impact of disease progression on the quality of life (QoL) of the caregiver at 6 and 12 months | baseline, 6 months, 12 months
  Caregiver QoL will be measured by the Parkinsonism Carers Quality of Life scale (PQoLCarers) (score range 0-104); higher score indicate worse QoL
To assess changes on the burden of orthostatic hypotension at 6 and 12 months from baseline | baseline, 6 months, 12 months
  Othostatic hypertension will be measured by the Orthostatic Hypotension Questionnaire (OHQ) (scores ranging from 0-100); higher scores indicate greater impairment
To describe occurrence of MSA subtypes and disease progression in each MSA subtype | baseline, 6 months, 12 months
  MSA subtype (i.e., MSA-P vs MSA-C) at each study site; disease progression will be measured by UMSARS
To assess the prevalence of "responders to Levodopa" (as per clinical judgement) at baseline and who continue to respond at 6 and 12 months from baseline | baseline, 6 months, 12 months
To describe Levodopa dose modifications from baseline to 6 and 12 months | baseline, 6 months, 12 months
To describe patient characteristics of responders to Levodopa versus non-responders to Levodopa, including: age (in years) at MSA onset, sex (male, female), MSA diagnosis (probable versus possible), MSA subtype (MSA-P versus MSA-C). | baseline, 6 months, 12 months
To characterise MSA symptoms and their progression over time | baseline, 6 months, 12 months
  MSA symptoms as per the following single items in UMSARS Part I (historical review):
  * Urinary incontinence (item 10)
  * Falling (item 8)
  * Speech (item 1)
  * Swallowing (item 2)
  * Walking (item 7)
To assess the psychometric properties of the Chinese version of UMSARS. | baseline, 6 months, 12 months
  To test the reliability and validity of the Chinese version of the UMSARS
To confirm the psychometric properties of the UMSARS | baseline, 6 months, 12 months
  To confirm the reliability and validity of the UMSARS Evaluation of UMSARS equivalence using Retrospective and Prospective Cohort data
To describe early MSA disease progression and mortality assessed remotely in 6-month intervals up until 60 months after enrolling in extension study. | 6-month intervals up until 60 months
  Disease progression in the extension will be assessed using:
  * UMSARS Part I
  * Mortality (date and cause of death)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (8):
- China (8):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing
  - Beijing Xuanwu Hospital, Capital Medical University, Beijing
  - Beijing Hospital, Beijing
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing
  - Xiangya Hospital of Central South University, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - Huashan Hospital of Fudan University, Shanghai
  - The Second Affiliated Hospital of Soochow University, Suzhou